CLINICAL TRIAL: NCT02442362
Title: Paclitaxel/Oxaliplatin/Fluorouracil (TOF) Regimen Versus S-1/Oxaliplatin (SOX) Regimen Metastatic Gastric Cancer Patients
Brief Title: TOF Versus SOX in Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Principal Investigator, Liangrong Shi, Director, The First People's Hospital of Changzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZ-GA-001
Record Dates: First submitted 2015-05-10; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TOF Group (Active Comparator): Patients in the TOF group received chemotherapy with "paclitaxel+oxaliplatin+fluorouracil"
  Interventions: Drug: paclitaxel+oxaliplatin+fluorouracil
- SOX Group (Experimental): The patients in the SOX group received chemotherapy with 'oxaliplatin+S1'
  Interventions: Drug: oxaliplatin+S1

INTERVENTIONS:
Drug: paclitaxel+oxaliplatin+fluorouracil — Patients treated with "paclitaxel+oxaliplatin+fluorouracil": paclitaxel (135 mg/m2 iv) on day 1, oxaliplatin (100 mg/m2 iv) on day 1, fluorouracil (500 mg/m2 continuous iv) on day 1-5twice/day for body surface area between 1.25 and 1.50 m2 orally) on days 1-14.
  Other Names: TOF regimen
  Arms: TOF Group
Drug: oxaliplatin+S1 — Patients treated with "oxaliplatin+S1": oxaliplatin (130 mg/m2 iv) on day 1 and S-1 (40 mg twice/day for body surface area < 1.25 m2 and 60 mg twice/day for body surface area between 1.25 and 1.50 m2 orally) on days 1-14
  Other Names: SOX regimen
  Arms: SOX Group

SUMMARY:
This study was designed to compare the efficacy and safety of aclitaxel/oxaliplatin/fluorouracil (TOF) regimen and S-1/oxaliplatin (SOX) regimen for metastatic gastric cancer (GC) patients.

DETAILED DESCRIPTION:
Gastric carcinoma ranks second among the most common causes of cancer deaths worldwide, with especial high prevalence in Asia . Gastric cancer is the third most common cancer in China and the incidence rate and death rate of gastric cancer in Jiangsu Province are especially higher than the national average. Surgical resection is the preferred treatment for gastric cancer, but approximately two-thirds of patients have metastatic disease at the time of diagnosis. Prognosis in these patients is poor, with a median survival time of 3 to 5 months without treatment and a reported 5-year survival rate of 9.4%. Even receiving curative gastrectomy, 60% of mGC patients develop local recurrences or distant metastasis.

For advanced-stage patients with inoperable gastric tumors, chemotherapy is considered the most effective treatment option and the efficacy of postoperative chemotherapy has been acknowledged. However, a worldwide consensus on standard chemotherapy regimens has yet to be established. The prognosis has gradually improved because of advances in chemotherapy regimens, but is not yet satisfactory.Among various regimens, the combinations of paclitaxel/oxaliplatin/fluorouracil (TOF) regimen and S-1/oxaliplatin (SOX) regimen have become two important ones.

Paclitaxel can bind to microtubules and induces hyperstabilization leading to cell cycle arrest and apoptosis. The response rate of GC patients to paclitaxel is 20%-25%. Oxaliplatin is a third-generation diaminocyclohexane platinum compound which has a wide range of antitumor activities, appearing to have a better safety profile than cisplatin. The response rate of mGC patients to FOLFOX-4 regimen is 38%-43%. S-1 is an oral anti-cancer agent composed of tegafur, 5-chloro-2,4-dihydroxypyridine, and oteracil potassium. The applying of S-1 as adjuvant chemotherapy for mGC can improve the overall survival (OS) and relapse-free survival. A meta-analysis showed OS favored S-1-based chemotherapy over 5-FU-based chemotherapy in mGC. S-1 plus oxaliplatin (SOX) have showed non-inferiority to S-1 plus cisplatin in PFS and that the treatment was well tolerated in patients with mGC.

No study is available comparing the efficacy and safety of TOF and SOX regimens. So the investigators performed the present randomized, controlled study to compare the efficacy and safety of the two regimens in mGC patients.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed mGC (stage IV)
2. ages between 20 and 80 years
3. measurable or assessable lesions by imaging studies according to the RECIST guideline 21
4. no prior chemotherapy except for postoperative adjuvant chemotherapy for more than 12 months before entry into the study
5. Eastern Cooperative Oncology Group (ECOG) performance status score less than 3
6. hepatic function

   * total bilirubin ≤ 1.5 × the institutional upper limit of normal value, aspartate aminotransferase/alanine aminotransferase ≤ 2.5 × the institutional upper limit of normal value, and alkaline phosphatase ≤ 2.5 × the institutional upper limit of normal value
   * renal function (serum creatinine level ≤ 1.5 mg/dL and creatinine clearance ≥ 50 ml/min)
   * adequate bone marrow function (hemoglobin level ≥ 90 g/L, white blood cell count of 4-10×109/L, neutrophil count ≥ 2×109/L, and platelet count ≥ 100×109/L)
7. estimated life expectancy more than 3 months
8. no other secondary malignant tumors.

Exclusion Criteria:

1. preexisted peripheral toxicity ≥ grade 2 of the National Cancer Institute Common Toxicity Criteria
2. concurrent or prior malignancy
3. central nervous system metastases
4. concurrent treatment that interfered with the study evaluation
5. active infection
6. other uncontrolled underlying medical conditions that would impair the ability of the patients to receive the planned treatment
7. having inadequate calorie and fluid intake
8. pregnant, and breastfeeding women or women of child-bearing potential without adequate contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Tumor respone | 8 weeks
  According to the RECIST guideline

SECONDARY OUTCOMES:
Side-effect | 8 weeks
  Safety was evaluated according to the NCI-CTC

CONTACTS AND LOCATIONS:
Overall Officials: Changping Wu, M.D., Study Director — the First People' Hospital of Changzhou